CLINICAL TRIAL: NCT06388733
Title: A Phase 3, Open-label, Randomized 2-arm Study Comparing the Clinical Efficacy and Safety of Niraparib With Temozolomide in Adult Participants With Newly-diagnosed, MGMT Unmethylated Glioblastoma
Brief Title: A Study Comparing Niraparib With Temozolomide in Adult Participants With Newly-diagnosed, MGMT Unmethylated Glioblastoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Ivy Brain Tumor Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: NeuroTrials, LLC (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IVY P3-24-021
Record Dates: First submitted 2024-04-24; First posted 2024-04-29 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-08

CONDITIONS: Glioblastoma; GBM; Brain Neoplasms, Adult, Malignant; Brain Tumor
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — niraparib; Temozolomide

STUDY DESIGN:
Masking Description: Blinded Independent Central Review is composed of independent radiologists and will be utilized to assess progression of disease
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Niraparib (Experimental)
  Interventions: Drug: Niraparib
- Arm B: Temozolomide (Active Comparator)
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: Niraparib — Participants will receive niraparib 200 mg orally once daily starting on Day 1 of RT. Following completion of RT, participants will continue niraparib adjuvant therapy orally once daily on Days 1 to 28 of each 28-day cycle until progression by BICR
  Other Names: Zejula
  Arms: Arm A: Niraparib
Drug: Temozolomide — Participants randomized to the comparator arm (Arm B) will receive SOC TMZ 75 mg/m2 orally once daily with RT starting on Day 1 of RT. Following completion of RT, participants will complete a 4-week rest period, and then receive adjuvant TMZ 150 to 200 mg/m2 orally once daily on Days 1 to 5 of each 28-day cycle until progression by BICR or for a maximum of 6 cycles.
  Other Names: Temodar; TMZ
  Arms: Arm B: Temozolomide

SUMMARY:
The goal of this Phase 3 clinical trial is to compare the efficacy of niraparib versus temozolomide (TMZ) in adult participants with newly-diagnosed, MGMT unmethylated glioblastoma multiforme (GBM). The main question it aims to answer is:

Does niraparib improve overall survival (OS) compared to TMZ?

Participants will be randomly assigned to one of two treatment arms: niraparib or TMZ.

* study drug (Niraparib) or
* comparator drug (Temozolomide - which is the standard approved treatment for MGMT unmethylated glioblastoma).

The study medication will be taken daily while receiving standard of care radiation therapy (RT) for 6-7 weeks.

Participants may continue to take the niraparib or TMZ adjuvantly as long as the cancer does not get worse or completion of 6 cycles of treatment (TMZ). A total of 450 participants will be enrolled in the study.

Participants' tasks will include:

* Complete study visits as scheduled
* Complete a diary to record study medication

ELIGIBILITY:
Inclusion Criteria:

* 1. Histologic documentation of a newly-diagnosed intracranial GBM, per 2021 WHO classification guidelines through local pathology review.
* 2. Age ≥18 years at the time of signing informed consent.
* 3. Sufficient tissue available for retrospective central pathology review, retrospective central confirmation of MGMT promoter methylation status and genomic analysis. If insufficient tissue is available,pproval may be granted on a case-by-case basis after a review.
* 4. Unmethylated MGMT promoter region determined locally by a validated PSQ or qMS-PCR assay compliant to local regulations. Numerical cut-off for an MGMT unmethylated tumor will be defined in the protocol.
* 5. Suitability for SOC RT to 60 Gy in 30 fractions using ESTRO-EANO 'single phase' targeting approach [Niyazi, 2023], per investigator's judgment.
* 6. No prior treatment for GBM (including brachytherapy or BCNU wafers), other than surgical resection or biopsy.
* 7. Female participants: Not pregnant, planning to get pregnant, or breastfeeding and one of the following conditions apply: is of nonchildbearing potential or is of childbearing potential AND using a contraceptive method that is highly effective (with a failure rate of <1% per year) from screening through at least 180 days after the last dose of study intervention. Breastfeeding is contraindicated during the study and for one month after the last dose of study intervention.
* 8. Male participants: Must agree to the following during the study intervention period and for at least 6 months after the last dose of study intervention: refrain from donation sperm PLUS be abstinent from heterosexual activity or agree to use a male condom and be advised of the benefit for a female partner to use a contraceptive method that is highly effective (with a failure rate of <1% per year).
* 9. The participant must be capable of providing signed informed consent, including compliance with the requirements and restrictions listed in the ICF and in this protocol.
* 10. Karnofsky performance status of ≥70.
* 11. Adequate organ function
* 12. Normal blood pressure (BP) or adequately treated and controlled hypertension (defined as systolic BP ≤140 mmHg and diastolic BP ≤90 mmHg).
* 13. Stable or decreased dose of dexamethasone, requiring no more than 5 mg daily equivalent dose, within 7 days before randomization.
* 14. Ability to swallow oral medications whole.

Exclusion Criteria:

* 1. Presence of metastatic or predominant leptomeningeal disease.
* 2. Current active pneumonitis or any history of pneumonitis requiring steroids (any dose) or immunomodulatory treatment within 90 days of planned start of the study.
* 3. Participant is at an increased bleeding risk due to concurrent conditions (e.g., major injuries or major surgery within the past 28 days prior to start of study treatment with the exception of tumor resection).
* 4. Any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach and/or bowels.
* 5. Has cirrhosis or current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal/gastric varices, or persistent jaundice. NOTE: Stable noncirrhotic chronic liver disease (including Gilbert's syndrome or asymptomatic gallstones), hepatobiliary involvement of malignancy, or chronic stable HBV infection (in a participant for whom HDV infection has been excluded) or chronic HCV infection is acceptable if the participant otherwise meets entry criteria.
* 6. Known human immunodeficiency virus (HIV) unless participants meet all of the following criteria:

  * Cluster of differentiation 4 ≥350/µL and viral load <400 copies/mL.
  * No history of acquired immunodeficiency syndrome-defining opportunistic infections within 12 months prior to enrollment.
  * No history of HIV-associated malignancy for the past 5 years.
  * Concurrent antiretroviral therapy as per the most current National Institutes of Health (NIH) Guidelines for the Use of Antiretroviral Agents in Adults and Adolescents Living with HIV [NIH, 2021] started >4 weeks prior to study enrollment.
* 7. MDS/AML or with features suggestive of MDS/AML.
* 8. History of another malignancy within 2 years prior to registration. Participants with a past history of adequately treated carcinoma-in-situ, basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or superficial transitional cell carcinoma of the bladder are eligible. Participants with a history of other malignancies are eligible if they have been treated with curative intent or continuously disease free for at least 2 years after definitive primary treatment.
* 9. Prior history of posterior reversible encephalopathy syndrome (PRES).
* 10. Any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study requirements and/or follow-up procedures.
* 11. Inability to undergo MRI brain with IV contrast.
* 12. Biopsy and/or resection (whichever is later) occurring >6 weeks prior to planned RT start date.
* 13. Surgical wound complication recovery at the time of enrollment.
* 14. Known hypersensitivity to the components of niraparib, TMZ, or their formulation excipients.
* 15. Known hypersensitivity to dacarbazine (DTIC).
* 16. Prior therapy with PARP inhibitors for systemic cancer.
* 17. Received a live vaccine within 30 days before the planned start of study intervention. Coronavirus disease 2019 (COVID-19) vaccines that do not contain live viruses are allowed. Note: mRNA and adenoviral-based COVID-19 vaccines are considered non-live.
* 18. Received a transfusion (platelets or red blood cells) or colony-stimulating factors (e.g., granulocyte macrophage colony-stimulating factor or recombinant erythropoietin) within 4 weeks of the planned start of study intervention.
* 19. Treatment with another investigational drug or other intervention within 5 half-lives of the investigational product.
* 20. Treatment with tumor treating fields (e.g., Optune) for GBM.
* 21. Presence of known isocitrate dehydrogenase (IDH) mutation.
* 22. Presence of known H3 mutation.
* 23. Previous diagnosis of WHO Grade 2 or 3 glioma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 24 months
  Overall survival, defined as the time from the date of randomization to the date of death due to any cause.

SECONDARY OUTCOMES:
Progression-free survival (PFS) assessed by Blinded Independent Central Review (BICR) | 24 months
  Progression-free survival, defined as the time from the date of randomization to the date of first disease progression per RANO 2.0 by BICR assessment or death from any cause, whichever occurs first.
Overall response rate | 24 months
  Percentage of patients who achieved confirmed complete response or confirmed partial response to treatment evaluated using RANO 2.0 by BICR.
Compare symptoms, function, and Health-related quality of life (HRQoL) and symptoms by EORTC QLQ-C30-item Core module (EORTC QLQ-C30) (Scores on a scale) | on Day 1 pre-dose or up to 7 days prior, on any day during the 6th week of RT, and on days of MRI at 4- and 12- weeks after RT, every 16 weeks thereafter on days of MRI
  EORTC QLQ-C30 is a validated questionnaire to assess overall health-related quality of life in participants with cancer.
Compare symptoms, function, and Health-related quality of life (HRQoL) and symptoms by EORTC QLQ-BN20-item Core module (EORTC QLQ-BN20) (Scores on a scale) | on Day 1 pre-dose or up to 7 days prior, on any day during the 6th week of RT, and on days of MRI at 4- and 12- weeks after RT, every 16 weeks thereafter on days of MRI
  EORTC QLQ-BN20 is a clinically valid and useful tool for assessing disease- and treatment-specific symptoms in brain neoplasm participants.
Compare symptoms, function, and Health-related quality of life (HRQoL) and symptoms by EQ-5D-3L | on Day 1 pre-dose or up to 7 days prior, on any day during the 6th week of RT, and on days of MRI at 4- and 12- weeks after RT, every 16 weeks thereafter on days of MRI
  The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
Changes from baseline in neurocognitive function assessed by Hopkins Verbal Learning test | on Day 1 pre-dose or up to 7 days prior, on any day during the 6th week of RT, and on days of MRI at 4- and 12- weeks after RT, every 16 weeks thereafter on days of MRI
  The Hopkins Verbal Learning Test is designed to evaluate memory. It requires participants to memorize a list of 12 items for 3 consecutive tests (recall), to identify the same 12 items from a list of semantically related or unrelated items (recognition), and to recall the same 12 items after a 15-minute delay (delayed recall).
Changes from baseline in neurocognitive function assessed by Controlled Oral Word Association | on Day 1 pre-dose or up to 7 days prior, on any day during the 6th week of RT, and on days of MRI at 4- and 12- weeks after RT, every 16 weeks thereafter on days of MRI
  The Controlled Oral Word Association Test is designed to evaluate verbal fluency. It requires participants to name words beginning with a specific letter with increasing associated activity, in 3 one-minute periods.
Changes from baseline in neurocognitive function assessed by Trail Making Test Parts A and B | on Day 1 pre-dose or up to 7 days prior, on any day during the 6th week of RT, and on days of MRI at 4- and 12- weeks after RT, every 16 weeks thereafter on days of MRI
  The Trail Making Test Part A is designed to evaluate visual motor scanning speed, and the Trail Making Test Part B is designed to evaluate executive function. These tests require participants to connect circles in numerical (Part A) or alternating numerical and alphabetical sequence (Part B) within a timed interval of less than 5 minutes for each test.
Incidence of participants with adverse events (AEs), serious adverse events (SAEs) and adverse events of special interest (AESIs) | 24 months
  AEs, SAEs and AESIs will be collected
Incidence of treatment discontinuations, dose interruptions, and dose reductions due to AEs, SAEs, or AESIs, changes in Karnofsky performance status, changes in clinical laboratory results, and vital sign measurements | 24 months
  Treatment discontinuations, dose interruptions, and dose reductions
Frequency and severity of symptomatic AEs based on PRO-CTCAE | 24 months
  The PRO-CTCAE is a patient-reported outcome measure developed to evaluate symptomatic toxicity in patients on cancer clinical trials.

CONTACTS AND LOCATIONS:
Overall Officials: Nader Sanai, MD, Study Chair — Ivy Brain Tumor Center
Locations (93):
- United States (30):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Ivy Brain Tumor Center, Phoenix, Arizona
  - Scripps Cancer Center, La Jolla, California
  - Moores UCSD Cancer Center, La Jolla, California
  - Indiana University, Indianapolis, Indiana
  - The NeuroMedical Center, Baton Rouge, Louisiana
  - MaineHealth Maine Medical Center Care, South Portland, Maine
  - Tufts Medical Center, Boston, Massachusetts
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Allina Health, Minneapolis, Minnesota
  - University of Minnesota Health Clinics and Surgery Center, Minneapolis, Minneapolis, Minnesota
  - Saint Lukes Neuro Oncology, Kansas City, Missouri
  - Washington University, School of Medicine, St Louis, Missouri
  - Atlantic Health System, Summit, New Jersey
  - Northwell Health, New Hyde Park, New York
  - New York University Ambulatory Care Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Duke Cancer Center Brain Tumor Clinic, Durham, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - University of Cincinnati Cancer Institute, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center Health System, Pittsburgh, Pennsylvania
  - Medical University of South Carolina - Department of Neurosurgery, Charleston, South Carolina
  - Baylor Scott & White Health, Temple, Texas
  - The University of Vermont Medical Center, Burlington, Vermont
  - University of Washington Medical Center, Seattle, Washington
  - University of Wisconsin Cancer Center, Madison, Wisconsin
- Australia (4):
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Austin Health, Heidelberg, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
- Canada (5):
  - BC Cancer - Vancouver, Vancouver, British Columbia
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network - Princess Margaret Cancer Centre, Toronto, Ontario
  - CHUM (Centre hospitalier de l'Université de Montréal), Montreal, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
- France (10):
  - CHU Nice - Hôpital Pasteur, Nice, Alpes Maritimes
  - Hôpital de la Timone, Marseille, Bouches-du-Rhône
  - Institut du Cancer de Montpellier, Montpellier, Herault
  - CRLCC Eugene Marquis, Rennes, Ille et Vilaine
  - ICO - Site René Gauducheau, Saint-Herblain, Loire Atlantique
  - Groupe Hospitalier Pitie-Salpetriere, Paris, Paris
  - Centre Hospitalier Universitaire de Lyon-Hospices Civils de Lyon-Hopital Pierre Wertheimer, Bron, Rhone
  - Centre Leon Berard, Lyon, Rhone
  - CHU Amiens-Picardie - Site Sud, Amiens, Somme
  - Centre Georges François Leclerc, Dijon
- Germany (8):
  - Universitaetsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Universitaetsmedizin Mannheim, Mannheim, Baden-Wurttemberg
  - Universitaetsklinikum Tuebingen, Tübingen, Baden-Wurttemberg
  - Universitaetsklinikum Regensburg, Regensburg, Bavaria
  - Universitaetsklinikum Bonn AoeR, Bonn, North Rhine-Westphalia
  - Klinikum Chemnitz gGmbH, Chemnitz, Saxony
  - Universitaetsklinikum Leipzig, Leipzig, Saxony
  - Vivantes Klinikum Neukoelln, Berlin, State of Berlin
- Italy (8):
  - IRCCS Istituto delle Scienze Neurologiche di Bologna, Bologna, Bologna
  - Azienda Ospedaliera Universitaria Careggi, Florence, Firenze
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Milano
  - Istituto Clinico Humanitas, Rozzano, Milano
  - A.S.L. Napoli 1 Centro Ospedale del Mare, Napoli, Napoli
  - IOV - Istituto Oncologico Veneto IRCCS, Padua, Padova
  - Azienda Ospedaliera Universitaria Policlinico Umberto I - Università di Roma La Sapienza, Rome, Roma
  - Azienda Ospedaliero-Universitaria Città della Salute e della Scienza di Torino, Torino, Torino
- Netherlands (2):
  - Maastricht UMC, Maastricht
  - UMC Utrecht, Utrecht
- Norway (2):
  - Oslo Universitetssykehus HF, Radiumhospitalet, Oslo
  - St. Olavs Hospital Hf, Universitetssykehuset i Trondheim, Trondheim
- Spain (12):
  - Hospital del Mar, Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona
  - Hospital Clinic de Barcelona, Barcelona, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba, Córdoba
  - ICO Girona - Hospital Universitari de Girona Dr Josep Trueta, Girona, Girona
  - Hospital Universitario Ramon y Cajal, Madrid, Madrid
  - Hospital Universitario 12 de Octubre, Madrid, Madrid
  - Hospital Universitario HM Madrid Sanchinarro, Madrid, Madrid
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Clinico Universitario de Salamanca, Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocio, Seville, Sevilla
  - ICO l'Hospitalet - Hospital Duran i Reynals, Barcelona
- Switzerland (4):
  - Universitaetsspital Basel, Basel
  - Ente Ospedaliero Cantonale, Bellinzona
  - Inselspital - Universitaetsspital Bern, Bern
  - Universitaetsspital Zürich, Zurich
- United Kingdom (8):
  - Bristol Haematology and Oncology Centre, Bristol, Avon
  - Addenbrooke's Hospital, Cambridge, Cambridgeshire
  - The Christie Hospital, Manchester, Greater Manchester
  - The Clatterbridge Cancer Centre, Metropolitan Borough of Wirral, Merseyside
  - Velindre Cancer Centre, Cardiff, South Glamorgan
  - Beatson West of Scotland Cancer Centre, Glasgow, Strathclyde
  - Queen Elizabeth Hospital, Birmingham, West Midlands
  - Guy's Hospital, London

IPD SHARING:
Plan to Share IPD: No